CLINICAL TRIAL: NCT04883125
Title: Potential Utility of Peroxisome Proliferator-activated Receptor Gamma Agonists in the Eradication of Chronic Myeloid Leukemia Stem Cells: Myth or Truth?
Brief Title: Value of Using Pioglitazone in Chronic Myeloid Leukemia Treatment
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Basma Atef, Assistant lecturer of Hematology (Internal medicine department), Mansoura University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MD/17.12.30
Record Dates: First submitted 2021-05-11; First posted 2021-05-12 (Actual); Last update posted 2021-05-12 (Actual); Status verified 2021-05

CONDITIONS: Chronic Myelogenous Leukemia, BCR-ABL Positive; CML, Chronic Phase
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Leukemia, Myeloid, Chronic-Phase | interventions — Pioglitazone; Imatinib Mesylate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Interventional no (Active Comparator): Patients treated with both drugs ( imatinib and pioglitazone)
  Interventions: Drug: Pioglitazone 15mg
- Control (No Intervention): Historical control (treated with imatinib only)

INTERVENTIONS:
Drug: Pioglitazone 15mg — pioglitazone (7.5-30 mg) once daily plus imatinib 400 mg 6 months
  Other Names: Imatinib 400mg
  Arms: Interventional no

SUMMARY:
Assessment of patients response and expression levels of CITED2 and HIF2a genes on adding pioglitazone to imatinib therapy.

DETAILED DESCRIPTION:
Eligible denovo CML patients will be treated by combination drug therapy of imatinib 400 mg plus pioglitazone (15 - 30mg).They will be on follow up for their complete blood count (CBC), chemistry profile and random blood sugar every 2 weeks. After 3, 6 and 12 months of treatment the patients response will be evaluated and compared with the obtained responses of a historical control group. Assessment of the hypoxia induced factor 2 alpha (HIF2a) gene and CBP/p300-interacting transactivator with glutamic acid (E) and aspartic acid (D)-rich tail 2 (CITED2) gene expression levels before and after 6 months of treatment will be additionally evaluated.

ELIGIBILITY:
Inclusion Criteria:

* CML cases (BCR-ABL1 positive)

Exclusion Criteria:

* Accelerated or blastic crisis
* Atypical CML (BCR-ABL1 negative)
* Chronic myelomonocytic leukemia (CMML)
* Pregnant or breastfeeding females.
* Patients with severe organ dysfunction

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2021-04-15 (Actual); Study Completion 2021-04-15 (Actual)

PRIMARY OUTCOMES:
Rate of major molecular response(MMR) at 12 months | 1 year
  Percentage of patients obtaining MMR at 12 months
Impact of treatment on the expression levels of stemness genes | 6 months
  Follow up the expression of CITED2 and HIF2a genes pattern

SECONDARY OUTCOMES:
Impact of treatment on the rate of transformation | 1 years
  Progression into accelerated or blastic phases

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed N. Mabed, Professor, Study Director — Oncology Center Mansoura University
Locations (1):
- Faculty of Medicine, Al Mansurah, Dakahlia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No